CLINICAL TRIAL: NCT06247969
Title: Using Cone Beam Computed Tomography For Appropriate Nostril Selection In Nasotracheal Intubation
Brief Title: Cone Beam Computed Tomography For Appropriate Nostril Selection for Nasotracheal Intubation
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, FUNDA ARUN, Assisstant Professor, Selcuk University
Other Study IDs: F001
Record Dates: First submitted 2024-01-20; First posted 2024-02-08 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Intubation; Difficult or Failed; Intubation Complication
Keywords: cone-beam computed tomography; intubation; nasal cavity; nasal septum; general anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients intubated under general anesthesia via nasotracheal route.: Patients intubated under general anesthesia via nasotracheal route successfully.
  Interventions: Device: endotracheal tube

INTERVENTIONS:
Device: endotracheal tube — Endotracheal Tube (ETT) is a flexible plastic tube that is inserted through the mouth or nose into the trachea to establish an artificial airway.

SUMMARY:
Design: Nasotracheal intubation is a standard blind procedure associated with various complications. Selection of the appropriate nostril is crucial in preventing most of these complications. The investigators aimed to evaluate the contribution of CBCT findings in selecting the proper nostril for nasotracheal intubation.

Methods: This prospective observational study outlines the protocol for research conducted at the Selçuk University Faculty of Dentistry.

Scope of the Research: The study encompasses patients undergoing dental surgery under general anesthesia at the Selçuk University Faculty of Dentistry.

1. Participant Selection: ASA I-II patients will be included in the study. Patients with structural abnormalities in the maxillo-mandibular anatomy, limited mouth opening, comorbidities such as rheumatoid arthritis, and a history of epistaxis will be excluded from the study.
2. Anesthesia Method: General anesthesia induction will be performed with intravenous (IV) propofol, IV rocuronium bromide, and IV fentanyl. Transition to nasotracheal intubation will follow adequate mask ventilation, and the preferred nostril will be determined through a simple occlusion test.
3. Data Collection: Demographic data, accompanying illnesses, medications used, and various parameters related to nasotracheal intubation will be recorded. The anesthetist performing nasotracheal intubation will be blinded to CBCT data, and the evaluation of data will be conducted jointly by the anesthetist and Radiology specialist after data collection from all patients is complete.
4. Exclusion Criteria: Unsuccessful nasotracheal intubation, difficult mask, and/or difficult intubation.
5. Implementation and Evaluation: Anesthesia procedures and CBCT evaluations will be carried out by experienced specialists.
6. The objective of this study is to evaluate the use of preoperative measurements of the nasal cavity from CBCT images in selecting the appropriate nostril for nasotracheal intubation under general anesthesia. The statistical tests to be employed are the chi-squared test and independent samples t-test.

DETAILED DESCRIPTION:
The goal of this prospective observational study is the contribution of CBCT findings in selecting the proper nostril for nasotracheal intubation. The main question it aim to answer is:

1. Can pre-operative evaluations of participiants' nasal cavity by using CBCT aid anesthetists for selecting the appropriate nostril for nasotracheal intubation? The participants will be informed both through a written consent form, and verbally that they would be participating in the observational study, and that apart from routine procedures, no additional interventions would be performed.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients

Exclusion Criteria:

* Clinical diagnosis of allergic rhinitis
* Patient with structural abnormalities in maxillo-mandibular anatomy,
* Patient with limited mouth opening
* Patient has previous history of epistaxis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population in this study consists ASA I-II patients, aged 18-70 years old, who had undergone maxillofacial surgery under general anesthesia with nasotracheal intubation and had undergone CBCT examination of maxillofacial area for various reasons before the operation.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Evaluation the use of preoperative measurements of the nasal cavity from CBCT images in selecting the appropriate nostril for nasotracheal intubation under general anesthesia. | 4 weeks
  The proper selection of the nostril is crucial in preventing complications such as bleeding associated with nasotracheal intubation. In this regard, we investigated the potential utility of Cone Beam Computed Tomography (CBCT), a commonly available imaging method in dental hospitals, as an assisting tool for anesthetists.

CONTACTS AND LOCATIONS:
Overall Officials: FUNDA ARUN, Principal Investigator — Selcuk University
Locations (1):
- Selcuk University Faculty of Dentistry, Konya, Turkey (Türkiye)